CLINICAL TRIAL: NCT00686920
Title: A Multi-Center, Open-Label Trial to Evaluate the Long-Term Safety and Tolerability of Rifaximin 550 mg BID in Subjects With a History of Hepatic Encephalopathy
Brief Title: Safety and Tolerability Study of Rifaximin in Participants With a History of Hepatic Encephalopathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RFHE3002
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-07

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rifaximin (Experimental): Participants from a previous rifaximin HE study and new participants were administered a single rifaximin 550 milligram (mg) tablet 2 times per day (approximately every 12 hours) for at least 24 months, until regulatory approval of rifaximin for reduction in risk of overt HE recurrence, or until the sponsor closed the study.
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Drug: Rifaximin — Oral
  Other Names: Xifaxan®

SUMMARY:
This study will look at the safety of a drug used in participants who have had hepatic encephalopathy (HE) in the past.

DETAILED DESCRIPTION:
Eligible participants had a history of HE, a Conn score of 0 to 2 at enrollment, and either had successfully participated in a previous HE study with rifaximin (that is, RFHE3001 [NCT00298038]), or were new participants enrolled with ≥1 verifiable episode of HE (equivalent to a Conn score of ≥2) associated with cirrhosis or portal hypertension within 12 months of screening.

Successful participation in a previous rifaximin study was defined as having received ≥80% and ≤120% of the expected tablets, having been reasonably compliant with study procedures, and having not been discontinued from the previous study due to study drug-related Adverse Events. Participants who experienced HE or associated symptoms during or after the RFHE3001 study were considered eligible for entry into this open-label study if the participant and Investigator did not perceive study medication as a possible cause of the HE episode or associated symptoms. Participants who did not participate in a previous HE study with rifaximin were eligible if this open-label study was the only rifaximin HE study available at an individual site.

ELIGIBILITY:
Inclusion Criteria:

* Must sign an Informed Consent Form
* In remission from past HE
* Appropriate birth control measures
* More than or equal to 18 years of age
* Must be potential for benefit from treatment
* Recent HE episodes
* Capable and willing to comply with all study procedures
* Participant has support network

Exclusion Criteria:

* Significant medical conditions or Investigator decision not to include the participant
* Allergies to the study drug or similar drugs
* Laboratory abnormalities
* Recent participation in another clinical trial
* Problems experienced in a previous HE trial
* Pregnant or at risk of pregnancy
* Recent alcohol consumption
* Active or latent bacterial or viral Infections
* Bowel issues
* Recent Active Cancer
* On a prohibited medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2007-03-07 (Actual); Primary Completion 2010-12-08 (Actual); Study Completion 2010-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Mathew, Study Director — Bausch Health Companies
Locations (35):
- United States (31):
  - Birmingham, Alabama
  - Aurora, California
  - Fresno, California
  - La Jolla, California
  - Long Beach, California
  - Los Angeles, California
  - Merced, California
  - Sacramento, California
  - San Francisco, California
  - Golden, Colorado
  - Washington D.C., District of Columbia
  - Macon, Georgia
  - Iowa City, Iowa
  - Monroe, Louisiana
  - Boston, Massachusetts
  - Detroit, Michigan
  - Kansas City, Missouri
  - Lebanon, New Hampshire
  - Bayside, New York
  - New York, New York
  - Rochester, New York
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - Odessa, Texas
  - San Antonio, Texas
  - Richmond, Virginia
  - Madison, Wisconsin
- Canada (4):
  - Calgary, Alberta
  - Victoria, British Columbia
  - Toronto, Ontario
  - Montreal, Quebec

REFERENCES:
- [Derived] Zacharias HD, Kamel F, Tan J, Kimer N, Gluud LL, Morgan MY. Rifaximin for prevention and treatment of hepatic encephalopathy in people with cirrhosis. Cochrane Database Syst Rev. 2023 Jul 19;7(7):CD011585. doi: 10.1002/14651858.CD011585.pub2. PMID 37467180
- [Derived] Mullen KD, Sanyal AJ, Bass NM, Poordad FF, Sheikh MY, Frederick RT, Bortey E, Forbes WP. Rifaximin is safe and well tolerated for long-term maintenance of remission from overt hepatic encephalopathy. Clin Gastroenterol Hepatol. 2014 Aug;12(8):1390-7.e2. doi: 10.1016/j.cgh.2013.12.021. Epub 2013 Dec 21. PMID 24365449

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 152 (47%) participants with hepatic encephalopathy (HE) rolled over from the double-blind study RFHE3001 (NCT00298038); 70 rifaximin participants (designated to the "Continued Rifaximin" arm in Study RFHE3002) and 82 placebo participants (designated to the "New Rifaximin" arm along with the new 170 [53%] participants in Study RFHE3002).
Groups:
- New Rifaximin: Participants new to receiving rifaximin were administered a single rifaximin 550 milligram (mg) tablet 2 times per day (approximately every 12 hours) for at least 24 months, until regulatory approval of rifaximin for reduction in risk of overt HE recurrence, or until the sponsor closed the study.
- Continuing Rifaximin: Participants who received rifaximin in the previous rifaximin HE study were administered a single rifaximin 550 milligram (mg) tablet 2 times per day (approximately every 12 hours) for at least 24 months, until regulatory approval of rifaximin for reduction in risk of overt HE recurrence, or until the sponsor closed the study.
Period: Overall Study
Arm/Group | New Rifaximin | Continuing Rifaximin
Started | 252 | 70
Received At Least 1 Dose Of Study Drug | 252 | 70
Completed | 120 | 34
Not Completed | 132 | 36
Not completed — Death | 45 | 14
Not completed — Liver Transplant | 23 | 8
Not completed — Recurrent Hepatic Encephalopathy Episode | 1 | 2
Not completed — Withdrawal by Subject | 23 | 5
Not completed — Protocol Violation | 2 | 1
Not completed — Adverse Event | 10 | 2
Not completed — Personal Reason | 0 | 1
Not completed — Lost to Follow-up | 15 | 3
Not completed — Moved to Another State | 1 | 0
Not completed — Transferred to Nursing Home | 1 | 0
Not completed — Noncompliance | 9 | 0
Not completed — Principal Investigator Decision | 2 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | New Rifaximin | Continuing Rifaximin | Total
Number analyzed (Participants) | 252 | 70 | 322
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (8.90) | 56.7 (9.36) | 57.4 (57.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 32 | 126
  Male | 158 | 38 | 196

OUTCOME MEASURES:

1. Secondary Outcome: Number Of Participants With Postbaseline Potentially Clinically Significant Laboratory (Hematology and Blood Chemistry) Abnormal Results In ≥5% of Participants
Description: Hematology and blood chemistry with potentially significant values included: Hemoglobin <9, >18, or ≥3 (grams/deciliter [g/dL]) decrease from previous visit or ≥4 g/dL decrease from baseline; Hematocrit <0.27%, >0.54%, or ≥0.10% decrease from previous visit or ≥0.15% decrease from baseline; Platelets <50 or >400*10^9/(liter [L]); Prothrombin time 9 seconds above baseline or upper limit of normal range; International normalized ratio >1.7; White blood cells <2.0 or >12.0*10^9/L; Lymphocytes <13.5% or >70%; Glucose, random, serum <2.2 or >16.5 millimole (mmol)/L; Potassium ≤3.0 or ≥5.5 mmol/L; Direct bilirubin increases 3-fold from baseline or >85.5 micromole (umol)/L. Baseline value was defined as the last available value (including the applicable values from the participants who rolled over from Study RFHE3001) prior to the first dose of study drug. A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline up to Month 36
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | New Rifaximin | Continuing Rifaximin
Number analyzed (Participants) | 252 | 70
Participants
  Hemoglobin: number analyzed (Participants) | 193 | 70
  Hemoglobin | 15 | 12
  Hematocrit: number analyzed (Participants) | 193 | 70
  Hematocrit | 12 | 4
  Platelets: number analyzed (Participants) | 193 | 70
  Platelets | 18 | 6
  Prothrombin Time: number analyzed (Participants) | 193 | 70
  Prothrombin Time | 16 | 7
  International Normalized Ratio: number analyzed (Participants) | 193 | 70
  International Normalized Ratio | 24 | 8
  White Blood Cells: number analyzed (Participants) | 193 | 70
  White Blood Cells | 15 | 2
  Lymphocytes: number analyzed (Participants) | 193 | 70
  Lymphocytes | 24 | 10
  Glucose, random, serum: number analyzed (Participants) | 193 | 70
  Glucose, random, serum | 8 | 8
  Potassium: number analyzed (Participants) | 193 | 70
  Potassium | 17 | 7
  Direct Bilirubin: number analyzed (Participants) | 193 | 70
  Direct Bilirubin | 14 | 5

2. Primary Outcome: Number Of Participants Reporting A Non-serious Adverse Event Or A Serious Adverse Event
Description: A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline up to Month 36
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | New Rifaximin | Continuing Rifaximin
Number analyzed (Participants) | 252 | 70
Participants
  Non-Serious Adverse Event | 78 | 15
  Serious Adverse Event | 158 | 49

3. Secondary Outcome: Number Of Participants With A Significant Mean Change From Baseline In Vital Signs
Description: Vital signs were measured and included sitting blood pressure, heart rate, oral temperature, and weight. These were collected at each scheduled study visit. Participants were placed supine for 5 minutes prior to each assessment of vital signs. Baseline value was defined as last available value (including the applicable values from the participants who rolled over from Study RFHE3001) prior to the first dose of study drug. A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline up to Month 36
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | New Rifaximin | Continuing Rifaximin
Number analyzed (Participants) | 252 | 70
Participants | 0 | 0

4. Secondary Outcome: Change From Baseline In Conn Score At Last Assessment
Description: The assessment for change in mental status during the study was measured by the Conn score (also known as the West Haven score). The following scale was used in the Conn scoring system: Grade 0=No personality or behavioral abnormality detected. Grade 1=Trivial lack of awareness, euphoria, or anxiety; shortened attention span; or impairment of addition or subtraction. Grade 2=Lethargy; disorientation for time; obvious personality change; and inappropriate behavior. Grade 3=Somnolence to semi-stupor, responsive to stimuli; confused; gross disorientation; and bizarre behavior. Grade 4=Coma, unable to test mental state. Participants entered the study with a Conn score of 0 to 2. Baseline value was defined as last available value (including the applicable values from the participants who rolled over from Study RFHE3001) prior to the first dose of study drug.
Time Frame: Baseline up to Month 36
Population: All participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | New Rifaximin | Continuing Rifaximin
Number analyzed (Participants) | 252 | 70
score on a scale
  Baseline | 0.4 (0.58) | 0.2 (0.40)
  Change from Baseline: number analyzed (Participants) | 246 | 70
  Change from Baseline | -0.1 (0.77) | 0.1 (0.41)

ADVERSE EVENTS:
Time Frame: Baseline up to Month 36
Description: All participants who received at least 1 dose of study drug.
Arm/Group | New Rifaximin | Continuing Rifaximin
Serious Adverse Events (participants affected / at risk) | 158/252 | 49/70
Other Adverse Events (participants affected / at risk) | 212/252 | 52/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | New Rifaximin (N=252) | Continuing Rifaximin (N=70)
Anaemia (Blood and lymphatic system disorders) | 19 | 6
Coagulopathy (Blood and lymphatic system disorders) | 2 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 1
Atrial flutter (Cardiac disorders) | 0 | 2
Cardiac arrest (Cardiac disorders) | 2 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 7 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 1
Mitral valve stenosis (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular hypokinesia (Cardiac disorders) | 1 | 0
Oculogyration (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 8 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Abdominal strangulated hernia (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 15 | 2
Colitis (Gastrointestinal disorders) | 1 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastroduodenal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 9 | 3
Haematemesis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 3 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Melaena (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 2
Oesophageal obstruction (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 4 | 3
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 9 | 2
Varices oesophageal (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2
Asthenia (General disorders) | 5 | 1
Chest pain (General disorders) | 4 | 0
Death (General disorders) | 1 | 0
Drug intolerance (General disorders) | 1 | 0
Generalised oedema (General disorders) | 2 | 2
Gravitational oedema (General disorders) | 1 | 0
Oedema (General disorders) | 3 | 0
Oedema peripheral (General disorders) | 3 | 1
Pyrexia (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Biliary cirrhosis primary (Hepatobiliary disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 7 | 7
Hepatic failure (Hepatobiliary disorders) | 23 | 5
Hepatic lesion (Hepatobiliary disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0
Hepatorenal failure (Hepatobiliary disorders) | 1 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 4 | 3
Liver disorder (Hepatobiliary disorders) | 5 | 0
Cryoglobulinaemia (Immune system disorders) | 1 | 0
Liver transplant rejection (Immune system disorders) | 0 | 1
Transplant rejection (Immune system disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 2 | 0
Biliary abscess (Infections and infestations) | 1 | 0
Biliary tract infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Campylobacter intestinal infection (Infections and infestations) | 0 | 1
Candida sepsis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 12 | 4
Cellulitis streptococcal (Infections and infestations) | 0 | 1
Central line infection (Infections and infestations) | 0 | 1
Clostridial infection (Infections and infestations) | 1 | 0
Clostridium colitis (Infections and infestations) | 3 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 2 | 0
Escherichia bacteraemia (Infections and infestations) | 2 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Fungal peritonitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Gastrointestinal candidiasis (Infections and infestations) | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 3 | 4
Meningitis cryptococcal (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 2 | 0
Peritonitis bacterial (Infections and infestations) | 9 | 1
Pneumococcal sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 13 | 3
Postoperative wound infection (Infections and infestations) | 1 | 0
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Scrotal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 7 | 1
Sepsis pasteurella (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 5 | 2
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 8 | 4
Urinary tract infection fungal (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 0 | 1
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Graft dysfunction (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Open wound (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Renal injury (Injury, poisoning and procedural complications) | 2 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Shunt stenosis (Injury, poisoning and procedural complications) | 1 | 0
Shunt thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Vena cava injury (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Ammonia increased (Investigations) | 2 | 0
Blood potassium decreased (Investigations) | 1 | 0
Central venous pressure decreased (Investigations) | 0 | 1
Transplant evaluation (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Haemochromatosis (Metabolism and nutrition disorders) | 1 | 0
Hyperammonaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 12 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 8 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 2
Liver carcinoma ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 2 | 0
Encephalopathy (Nervous system disorders) | 2 | 1
Hepatic encephalopathy (Nervous system disorders) | 79 | 18
Mental impairment (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Aggression (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 12 | 2
Renal failure acute (Renal and urinary disorders) | 30 | 5
Renal failure chronic (Renal and urinary disorders) | 1 | 2
Renal impairment (Renal and urinary disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hepatopulmonary syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Penile ulceration (Skin and subcutaneous tissue disorders) | 1/158 | 0/38 — This is a sex-specific adverse event that only affects male participants.
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Liver transplant (Surgical and medical procedures) | 22 | 7
Renal transplant (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0
Peripheral occlusive disease (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 2 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | New Rifaximin (N=252) | Continuing Rifaximin (N=70)
Anaemia (Blood and lymphatic system disorders) | 28 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 4
Nausea (Gastrointestinal disorders) | 52 | 15
Ascites (Gastrointestinal disorders) | 38 | 6
Vomiting (Gastrointestinal disorders) | 34 | 8
Abdominal pain (Gastrointestinal disorders) | 30 | 8
Diarrhoea (Gastrointestinal disorders) | 29 | 9
Constipation (Gastrointestinal disorders) | 33 | 4
Abdominal pain upper (Gastrointestinal disorders) | 15 | 5
Varices oesophageal (Gastrointestinal disorders) | 13 | 7
Haemorrhoids (Gastrointestinal disorders) | 9 | 4
Oedema peripheral (General disorders) | 48 | 13
Fatigue (General disorders) | 31 | 7
Pyrexia (General disorders) | 14 | 6
Oedema (General disorders) | 17 | 2
Asthenia (General disorders) | 14 | 3
Cholelithiasis (Hepatobiliary disorders) | 9 | 4
Urinary tract infection (Infections and infestations) | 50 | 15
Upper respiratory tract infection (Infections and infestations) | 15 | 4
Cellulitis (Infections and infestations) | 16 | 1
Pneumonia (Infections and infestations) | 15 | 2
Peritonitis bacterial (Infections and infestations) | 6 | 4
Procedural pain (Injury, poisoning and procedural complications) | 16 | 3
Contusion (Injury, poisoning and procedural complications) | 8 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 37 | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 15 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 15 | 5
Dehydration (Metabolism and nutrition disorders) | 13 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 13 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 10 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 30 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 23 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 4
Dizziness (Nervous system disorders) | 25 | 7
Headache (Nervous system disorders) | 22 | 5
Depression (Psychiatric disorders) | 30 | 9
Insomnia (Psychiatric disorders) | 30 | 4
Anxiety (Psychiatric disorders) | 15 | 8
Renal failure acute (Renal and urinary disorders) | 13 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 14 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 20 | 3
Rash (Skin and subcutaneous tissue disorders) | 19 | 4
Hypotension (Vascular disorders) | 17 | 4
Hypertension (Vascular disorders) | 16 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.